CLINICAL TRIAL: NCT03719872
Title: Utility of Bedside Ultrasound for Diagnosis of Intraperitoneal Free Air
Brief Title: Point of Care Ultrasound for Diagnosis of Abdominal Free Air
Status: Completed | Type: Observational
Sponsor: David Blehar (Other)
Responsible Party: Sponsor-Investigator, David Blehar, Associate Professor of Emergency Medicine, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Other Study IDs: H-00013680
Record Dates: First submitted 2018-10-19; First posted 2018-10-25 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Free Air in Abdomen
Keywords: laparoscopic surgery; transabdominal ultrasound; Free air
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Participants undergoing laparoscopy: Participants undergoing laparoscopic abdominal surgery with surgical insufflation receiving pre-operative transabdominal ultrasound and post-operative transabdominal ultrasound.
  Interventions: Diagnostic Test: Pre-Operative Transabdominal Ultrasound; Diagnostic Test: Post-Operative Transabdominal Ultrasound

INTERVENTIONS:
Diagnostic Test: Pre-Operative Transabdominal Ultrasound — Pre-Operative Transabdominal Ultrasound evaluation of the right upper quadrant of the abdomen. Examination with be performed with low frequency curvilinear transducer and high frequency linear transducer at 5 standardized locations along the right costal margin followed by a 10 second sweep along the costal margin from the xyphoid process to the mid-axillary line
Diagnostic Test: Post-Operative Transabdominal Ultrasound — Post-Operative Transabdominal Ultrasound evaluation of the right upper quadrant of the abdomen. Examination with be performed with low frequency curvilinear transducer and high frequency linear transducer at 5 standardized locations along the right costal margin followed by a 10 second sweep along the costal margin from the xyphoid process to the mid-axillary line

SUMMARY:
This study evaluates the ability of ultrasound to identify intraperitoneal free air. The study will consist of blinded review of abdominal ultrasound images of patients before and after laparoscopic surgery, a procedure which results in the introduction of air into the peritoneal cavity.

DETAILED DESCRIPTION:
Free peritoneal air is a marker of potential intraabdominal catastrophe, reflecting perforation of a hollow viscous organ such as stomach or intestine. While definitively identified by computed tomography, this diagnostic test can be delayed. Presence of air beneath the diaphragm on an upright chest or abdominal radiograph can allow for faster diagnosis, but again can present limitations in terms of timing.

Bedside clinician performed ultrasound has become standard practice in emergency medicine and critical care settings. Traditionally, air is not conducive to diagnostic ultrasound, but the artifacts it creates can be used to give clues about certain conditions. Recently this artifact has been proposed as a means to identify free peritoneal air. Several small studies have shown promise for the technique, but further investigation is warranted.

In this study the investigators will generate a database of standardized abdominal ultrasound images in subjects undergoing laparoscopic surgery. During this surgery, the peritoneal cavity is intentionally insufflated with air. The majority of this is removed at the end of the case, but small volumes of air remain, as evidence by the presence of air on CT scan when performed shortly after surgery.

The investigators will obtain a standardized set of images preoperatively and post operatively which will then be reviewed in a blinded fashion by three expert reviewers, one each from radiology, surgery and emergency medicine, with data analysis to determine sensitivity and specificity of ultrasound for free air.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled for elective laparoscopic surgery
* Age 18 or greater

Exclusion Criteria:

* Age less than 18
* Pregnant
* unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects drawn from population of surgical patients at UMassMemorial Medical center undergoing elective laparoscopic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Presence of Free Air Artifact on Ultrasound | Following completion of laparoscopic surgery, average of 2 hours, up to 1 day.
  Hyperechoic echo originating from peritoneal stripe

CONTACTS AND LOCATIONS:
Overall Officials: David Blehar, MD, Principal Investigator — UMASS MEDICAL SCHOOL
Locations (1):
- UMass Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No